CLINICAL TRIAL: NCT06823115
Title: Assessment of Worldwide Acute Kidney Injury Epidemiology in Neonates 2.0: Towards Expanding Our Understanding of Neonatal Acute Kidney Injury
Brief Title: Assessment of Worldwide Acute Kidney Injury Epidemiology in Neonates 2.0
Acronym: AWAKEN 2
Status: Enrolling by invitation | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Neonatal Kidney Collaborative (Unknown)
Responsible Party: Principal Investigator, Michelle Casey Starr, Assistant Professor oof Pediatrics, Indiana University
Other Study IDs: 23847
Record Dates: First submitted 2025-02-04; First posted 2025-02-12 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury; Fluid Overload; Prematurity Complications; Risk Factors; Epidemiology; Chronic Kidney Disease(CKD); Hypertension
Keywords: acute kidney injury; chronic kidney disease; neonates; prematurity; hypertension
MeSH Terms: conditions — Acute Kidney Injury; Edema; Renal Insufficiency, Chronic; Hypertension; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Neonates at Risk of Kidney Disease: Inclusion Criteria
  1. Admitted to participating NICUs between 1/1/19- 3/31/19
  2. > 48 hours of IV fluids
  Exclusion Criteria
  1. Age > 14 days at admission
  2. Congenital heart disease requiring transfer for escalation of CHD care and/or surgery within the first 7 days
  3. Lethal chromosomal anomalies
  4. Neonatal mortality <48 hours

SUMMARY:
There is a growing focus on short- and long-term kidney health in neonates, including those with acute kidney injury (AKI). AKI occurs commonly in the Neonatal Intensive Care Unit (NICU) and is associated with adverse outcomes. In addition to poor outcomes during the hospitalization, infants discharged from the NICU may have an increased burden of kidney disease during childhood. Studies of long-term kidney function in children born prematurely show a fourfold increase in chronic kidney disease (CKD) by adolescence and into adulthood.

Despite the landmark findings of the Assessment of Worldwide Acute Kidney Injury Epidemiology in Neonates (AWAKEN) study, the limitations of this study are notable. First, the AWAKEN study enrolled infants admitted in 2014, making the data now over 10 years old. Much has changed in neonatal practice (e.g. increased AKI awareness, treatment strategies). Secondly, the findings of the AWAKEN study were geographically limited. While the AWAKEN study was multi-national and multi-center, it represented only 24 centers (22 from North America, 1 from India and 1 from Australia). Finally, information collected from AWAKEN ended at hospital discharge.

The investigators seek to leverage the strength of the Neonatal Kidney Collaborative along with other organizations and collaboratives interested in neonatal kidney health to address these gaps. Therefore, the investigators are conducting a second, modified iteration of this study entitled "AWAKEN 2.0". AWAKEN 2.0 will be a multi-center multi-national retrospective analysis utilizing similar methodology to the AWAKEN study.

DETAILED DESCRIPTION:
AWAKEN 2.0 is a multi-center multi-national retrospective analysis utilizing similar methodology to the AWAKEN study. The investigators will capture information on all infants admitted to participating level 3 and 4 NICUs between January 1-March 31, 2019, to answer specific hypothesis regarding the following three inter-connected but independent specific aims:

Specific Aim 1. Describe prevalence of AKI in a multi-national multi-center retrospective cohort, 5 years after the original AWAKEN study.

1. Primary hypothesis: The investigators hypothesize that rates of neonatal AKI are higher than the rate described in the original AWAKEN study.
2. Population:

   1. Inclusion Criteria include all infants admitted to participating NICUs between 1/1/19- 3/31/19 and receiving > 48 hours of IV fluids
   2. Exclusion Criteria include age > 14 days at admission, congenital heart disease requiring transfer for escalation of CHD care and/or surgery within the first 7 days, lethal chromosomal anomalies and/or neonatal mortality <48 hours
3. Primary Outcome - Neonatal AKI
4. Potential confounders - gestational age, birth weight, 5 minute APGAR score, multiple gestation, significant renal anomalies, site characteristics.

Specific Aim 2. Determine if AKI is independently associated with mortality, length of stay, and discharge serum creatinine (SCr).

1. The investigators hypothesize that higher stages of AKI are associated with higher mortality, longer lengths of stay and higher serum creatinine at discharge, even after controlling for confounding factors.
2. Populations - Same as Specific Aim 1.
3. Primary Exposure - Neonatal AKI definitions (table 3)
4. Primary Outcome - Survival
5. Secondary outcomes will include: Hospital length of stay, BPD.
6. Potential confounders - gestational age, birth weight, 5 minute APGAR score, multiple gestation, significant renal anomalies,
7. Exploratory outcomes - recognize that the proposed definition may not be the best definition to predict clinical outcomes. Also recognize that there may be a need to have different definitions for premature infants. The investigators plan to explore how other definitions reported in the literature can predict these outcomes (for example using the 90th % for normative values). In addition, this will have the largest comprehensive database to explore new definitions which could incorporate fluid balance and other factors.

Specific Aim 3. Determine if AKI can predict chronic kidney disease, recurrent AKI and hypertension during early childhood.

1. The investigators hypothesize that higher stages of AKI are associated with chronic kidney disease and recurrent AKI during early childhood.
2. Population - Same as Specific Aim 1
3. Primary Exposure - Neonatal AKI definitions (table 3)
4. Primary Outcome - Childhood CKD
5. Secondary Outcomes - Childhood hypertension, recurrent AKI and childhood ESRD.

Each participating site will screen all neonates admitted to the NICU during the 3 months of study and capture additional data on those who meet the same inclusion and exclusion criteria as the original cohort. There will be 6 different integrated forms.

1. Screening form (all infants)
2. Baseline form for included infants (maternal demographic data, admission indication)
3. First 14 days form (i.e. urine output, medications and respiratory support)
4. Serum creatinine data (all values from date of birth to date of IRB approval)
5. Discharge form (discharge diagnoses, medications, follow-up anticipated)
6. Follow-up Information (clinically obtained follow-up after discharge)

ELIGIBILITY:
Inclusion Criteria:

1. All infants born or admitted to a participating level 3 or 4 NICU between 1/1/19- 3/31/19 will be screened.
2. Infants who received intravenous fluids for > 48 hours will be eligible.

Exclusion Criteria:

1. Age > 14 days at admission
2. Congenital heart disease requiring transfer for escalation of CHD care and/or surgery within the first 7 days
3. Lethal chromosomal anomalies
4. Neonatal mortality <48 hours

Ages: 0 Minutes to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The investigators will conduct a multi-center retrospective cohort study. All infants admitted to the NICU between January 1, 2019 and March 31, 2019 will be screened for the study.The investigators will enroll eligible infants who meet inclusion and exclusion criteria at each center for 3 consecutive months. Based on average admissions for 2018 at our centers who meet inclusion and exclusion criteria, it is estimated that it can enroll approximately 4000 infants during this time.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Neonatal Acute Kidney Injury | Up to 6 months or NICU discharge, whichever comes first
  The investigators will evaluate the rate of neonatal AKI among infants that meet inclusion criteria across all sites. Neonatal Acute Kidney Injury will be defined by the standard neonatal definitions, including serum creatinine values and urine output (when available). Furthermore, investigators will examine if different thresholds or definitions of AKI will better predict outcomes.

SECONDARY OUTCOMES:
Risk factors for Neonatal AKI | Up to 6 months or NICU discharge, whichever comes first
  Define the major risk factors associated with neonatal AKI. The investigators will randomly split the cohort into two groups. The investigators will develop a risk factor prediction model with the first group, and test the ability of the model to predict AKI with the second group.
Fluid Overload | NICU admission through discharge.
  Fluid overload will be calculated based on daily weights and intake and output values. We will determine how fluid balance during the first few weeks of life relates to biochemical data and clinical outcomes.
Mortality | Up to 6 months or NICU discharge, whichever comes first
  Determine if the KDIGO AKI definition adapted to neonates can predict mortality. Investigators will also evaluate if other thresholds or proposed AKI definitions can better predict mortality.
Chronic Kidney Disease | NICU discharge to 5 year follow-up
  In infants with available follow-up data clinically obtained, investigators will determine the rates of both clinically diagnosed (by ICD code or note) and laboratory determined Chronic Kidney Disease (using the CKID-U25 eGFR definitions).
Hypertension | NICU discharge to 5 year follow-up
  In infants with available follow-up data clinically obtained, investigators will determine the rates of both clinically diagnosed (by ICD code or note) and value determined hypertension (using AAP Hypertension thresholds)
Proteinuria | NICU discharge to 5 year follow-up
  In infants with available follow-up data clinically obtained, investigators will determine the rates of both clinically diagnosed (by ICD code or note) and laboratory determined proteinuria.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
As a retrospective study and based on terms of the data sharing agreements between sites, individual patient level data will not be made available. Investigators that have questions that may be answered by the data will be able to present proposal to request secondary data analyses to be conducted on de-identified data.